CLINICAL TRIAL: NCT03600025
Title: Investigation of Innate Immune Responses to Salmonella Typhi in Typhoid Fever in Children and Adults Patients and Vaccinees in Dhaka, Bangladesh
Brief Title: Cellular Immune Responses in Typhoid Fever Patients and Vaccinees
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR-17082
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-07

CONDITIONS: Typhoid Fever Patients and Healthy Volunteers to Receive Typbar-TCV Vaccine

STUDY DESIGN:
Intervention Model Description: Apparently healthy volunteers will receive typhoid vaccine one time point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-randomized (Other): Responses will be compared before and after vaccination
  Interventions: Biological: Typbar-TCV vaccine

INTERVENTIONS:
Biological: Typbar-TCV vaccine — vaccine will receive intramuscularly

SUMMARY:
Typhoid fever caused by Salmonella Typhi and Paratyphi causes over 21 million cases of febrile illness and 200,000 deaths are attributed to enteric fever each year. Typhoid fever is an enteric infection that results in febrile illness. Typhoid fever causes significant morbidity in the developing world especially young children.S. Typhi specific antibody responses are elicited in typhoid fever and following typhoid vaccination. Cross-reactive multifunctional CD+4 T cell mediated IL-17 responses have been shown in typhoid fever. As S. Typhi as an intracellular pathogen, cellular immune responses might be central to protection. S. Typhi peptide subunit vaccine elicits CD+4 T cell responses that correlate with protection in mice. The role of mucosal associated invariant T cell (MAIT) and natural killer (NK) cell responses in typhoid fever or following vaccination remain poorly understood. Transcriptome profiling of human immune responses to S. Typhi infection is not clearly understood. Establishing successful infection by S. Typhi evasion of T cell and neutrophil responses need to be investigated to better understand the correlates of protection.

DETAILED DESCRIPTION:
Description of the Research Project: It has been previously shown that IFN-gamma and IL-17 are increased in typhoid fever patients. It was shown that S. Typhi infection induces antibody responses against a number of key typhoid antigens (LPS) HlyE, Flagellar protein FliC and chaperon protein EcpD). In the enteric diarrheal disease cholera, MAIT cells are activated and associated LPS specific antibody responses are generated. In a human challenge model study, it has been shown that CD8+ T cell memory cells are key correlates of protection against typhoid fever. The live attenuated typhoid vaccine (TY21a) also induces MAIT cells after immunization. It has been shown that IL-12, IL-15, IL-18 induce memory-like NK cells in a mouse model and IL-21 induces memory-like NK cells protective against Mycobacterium tuberculosis infection. The role of activated MAIT cells, and cytokine induced memory-like NK cells in typhoid fever currently unknown.

One of the multiple killing mechanism employed by neutrophil is the release of neutrophil extracellular traps (NETs) that contain myeloperoxidase (MPO), elastase, lysozyme and defensins. Infection induces releases of NETs to trap microbial pathogens. Neutrophils isolated from typhoid fever patients release NETs in and that neutrophil NET release is primed by vaccination with a subunit-conjugate vaccine.

Study intervention: Typbar-TCV is a Typhoid Vi capsular polysaccharide tetanus toxoid conjugate vaccine. Typbar-TCV is the world's 1st clinically proven conjugate typhoid vaccine. This vaccine is WHO pre-qualified and approved for children and infants less that 2 years of age. During the Phase III clinical study, a single dose of Typbar-TCV elicited 4-fold seroconversion rates of 98.05%, 99.17% and 92.13% in subjects between greater than 6 months to 2 years, >2 to 15 years and >15 to 45 years respectively. Each volunteer in the vaccination arm of the study will receive 25 ug of Typbar-TCV vaccine administered as 0.5 ml single intracellular dose.

Storage condition: The vaccine will be stored at +2-8C and cold chain will be maintained at all times.

Study participants and sample collection: The investigators will collect 8-10 ml of blood from adults and 3-5 ml of blood from children who will be suspected typhoid fever patients (age 1-59 years) at enrollment (day1) and if patient is S. Typhi/Paratyphi culture confirmed then two more blood samples (2-5 days and 27-33 days later) will be collected. The investigators will collect 8-10 ml of blood from adults and 3-5 ml of blood from children before vaccination (day 0) and two more blood samples after one dose of vaccination at day 7 (6-8 days later) [13] and at day 30 (27-33 days later). Peripheral blood mononuclear cells (PBMCs) and neutrophils will be isolated from blood samples and will be used for different assays (Polymorphprep kit). Plasma samples will be separated to measure antibody response to infection and vaccination.

Patient management Depending on discretion of clinician, treatment of the patient with antibiotic and other necessary drug will be provided. After culture confirmation of typhoid fever antibiotic treatment will be adjusted depending on antibiotic sensitivity pattern. If patient does not respond to oral antibiotic then we will provide injectable antibiotic. If the patient remains unresponded to injectable antibiotic and/or other complication arise, then the patient will be hospitalized. The investigators are conducting another typhoid study where the patients are enrolled in different health care facilities in Mirpur and also icddr,b Dhaka hospital. The patient management will be supported by other ongoing typhoid project.

Laboratory Assay Procedure:

MAIT and NK cell assay: Isolated PBMCs will be stained with fluorochrome labelled antibodies and flow cytometric phenotyping performed (acquisition of ≥50000 live cells on a FACS-Aria). MAIT cells will be defined as live (DAPI-) CD3+CD4-CD161hiVα7.2+ cells, expressed as a percentage of total CD3+ lymphocytes, and CD38 used as a marker of cell activation. The investigators will also assess the frequency of circulating live CD3+CD8+CD4-CD161loVα7.2+ cells, which have been suggested to be MAIT-derived cells associated with absent or reduced cytokine secretion in vitro. CD4+ (live CD3+ CD8-CD4+) T cell responses in study subjects will be evaluated in different T memory (TM) subsets defined by their expression of CD45RA and CD62L i.e., T central memory (TCM; CD45RA-CD62L+), T effector memory (TEM; CD45RA-CD62L-) and T effector memory CD45RA+ (TEMRA; CD45RA+CD62L-), T follicular (CD3+CXCR5+) and Naïve T cells (TN: CD45RA+CD62L+). Activated NK cell as live CD3-, CD45+, CD56+, CD69+, CD40L+, CD16+ cells and memory like NK cell as live CD3-CD56+CD16+NKp46+CD27+.

Cytokine analysis: Isolated lymphocytes will be stimulated with S. Typhi antigens (Whole cell, MP and LPS) for 48 hours as well as for 5 days and culture supernatant will be collected and stored until analyzed at -70°C. Cytokines in culture supernatant will be analyzed by using multiplex bead array (Luminex).

Quantitation of NETs: Neutrophils will be isolated from peripheral blood based on previously described method. The release of NETs will be measured by neutrophil NET assay kit (NET assay kit, Creative Biomart, NY, USA). NETosis will be quantified by measuring levels of elastase that are released from neutrophils and NETs mediated killing will be quantified by measuring viability of bacteria.

NETs mediated killing assay: To determine the efficiency of NETs in killing S. Typhi, a CFU assay will be performed. Overnight culture S. Typhi will be co-incubated with freshly isolated human neutrophils in 96-well culture plate and incubated at 37ºC. After 3 hours of incubation, wells will be aspirated and washed with PBS. Dilutions of 1:10 and 1:100 will be made and 100 µl of each dilution will be plated onto Brain Heart Infusion (BHI) agar. Culture plates will be incubated at 37ºC with 5% CO2. The number of CFU will be counted after 24 hours incubation and after 3 days of culturing until no further increase in colony numbers are observed.

Neutrophil intracellular metabolite assay: Neutrophils will be isolated from blood and incubated at 37ºC for 1 hour for recovery. Incubation media will be aspirated and 1 ml of dry ice (-80ºC) cold 80% methanol will be added. Cells will be vortexed for 1 min, and then centrifuged at 15 K rpm for 1 min. Supernatant will be collected in tubes and stored at -80ºC until use. Before analysis samples will be removed from -80ºC and allow to equilibrate to room temperature. Supernatant (75 µl) will be transferred to a liquid chromatography-tandem mass spectrometry (LC-MS) vial capped. Ten microliters of sample will be autoloaded into LC-MS system for metabolite separation and mass spectrometric analysis.

Antibody responses to lipopolysaccharide (LPS) in plasma. Plasma antibody responses to S. Typhi LPS in patients and vaccinees will be measured using ELISA methods. Briefly, 96-well microtiter plates will be coated with LPS and incubated with plasma (1:10 dilution) with serial 3-fold dilutions thereafter. Plates will be washed, and horseradish peroxidase-conjugated anti-human IgA, IgG and IgM antibodies will be added. Plates will be developed using 0.1% ortho-phenylene diamine (OPD) and 0.1% hydrogen peroxide (H2O2), and OD will be measured at 492 nm. A 2-fold or higher antibody response will be considered a significant response.

Transcriptomics analysis: From a subset of adult patients and vaccinees 3 ml blood will be collected in Tempus RNA tubes (applied biosystem) and RNA will be extracted from blood, trancriptomic sequencing will be done at Shanghi, China (BGI) which is a service providing lab and data will be analyzed using next-gen RNA-seq sequencing to see the gene expression profile. Differential gene expression will be analysed using the DESeq package (Bioconductor). The obtained sequence reads will be normalized between patients/vaccinees versus healthy controls. A ratio larger than 2 and lower that 0.5 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria 1. Apparently healthy

Exclusion Criteria:

* 1. Previously history of illness in the last one month. 2. History of taking typhoid vaccine and history of typhoid fever. 3. History of taking any other live or killed enteric vaccine in the last 4 weeks.

Ages: 1 Year to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
MAIT cells and NK cells in the typhoid vaccine recipients | up to 30 days
Roles of IL-21, IL-12. IL-15 and IL-18 in the activation of natural killer cells and generation of memory like NK cells in typhoid fever and vaccinees | up to 30 days
In vitro capacity of NETs to trap and kill S. Typhi | up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrheal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No